CLINICAL TRIAL: NCT01732068
Title: Phase II Study for the Treatment of Poor Ovarian Responders With Corifollitropin Alfa Followed by hpHMG in a Short GnRH Agonist Protocol
Brief Title: Treatment of Poor Ovarian Responders With Corifollitropin Alfa Followed by hpHMG in a Short GnRH Agonist Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nikolaos P. Polyzos, Principal investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/082
Record Dates: First submitted 2012-11-17; First posted 2012-11-22 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Infertility; Poor Ovarian Response
Keywords: Poor ovarian response; Poor ovarian responders; Bologna criteria for poor ovarian response
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Corifollitropin alfa+hMG (Experimental)
  Interventions: Drug: Triptorelin; Drug: Corifollitropin alfa; Drug: hpHMG

INTERVENTIONS:
Drug: Triptorelin — Triptorelin 0.1 mg/1 ml solution daily from day 1 or 2 of the cycle onwards
Drug: Corifollitropin alfa — Corifollitropin alfa 150μg (single dose) on day 2 or 3 of the cycle
Drug: hpHMG — 300IU hMG daily from day 7 following Corifollitropin alfa until the day of ovulation triggering

SUMMARY:
The purpose of the present study is to examine the level of ovarian response and the pregnancy rates among poor ovarian responders treated with a novel treatment protocol with 150μg corifollitropin alfa followed by 300IU hMG in a short GnRH agonist protocol.

DETAILED DESCRIPTION:
Corifollitropin alfa reaches maximum concentrations (Cmax), between 25 and 45 h after injection , a time interval which is significantly shorter as compared to treatment with rFSH. The investigators hypothesized that this rapid increase in the serum FSH concentration may result in a significantly higher exposure of the small antral follicles to constant high levels of FSH during the early follicular phase, securing not only the recruitment of the follicles, but also the continued growth.

In the current study the investigators examine whether administration of corifollitropin followed by 300IU hMG in a short GnRH agonist protocol may result in acceptable pregnancy rates in poor ovarian responders fulfilling the "Bologna criteria"

ELIGIBILITY:
Inclusion Criteria:

Patients should fulfill the "Bologna criteria" for poor ovarian response

At least two of the following three features must be present:

i. Advanced maternal age (≥40 years) or any other risk factor for POR (poor ovarian response); ii. A previous POR (≤3 oocytes with a conventional stimulation protocol); iii. An abnormal ovarian reserve test (i.e. AFC <7 follicles or AMH <1.1 ng/ml).

Two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ORT (ovarian reserve test).

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10 to 12 weeks of gestation

SECONDARY OUTCOMES:
Number of oocytes retrieved | Day of oocyte retrieval
Cycles with embryo transfer | Day of Embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Centre for Reproductive Medicine UZ Brussel, Brussels, Belgium